CLINICAL TRIAL: NCT01887951
Title: Clinical Evaluation of Penthrox (Methoxyflurane)and Tramadol for the Singapore Emergency Ambulance Service
Brief Title: Penthrox Versus Tramadol for SCDF
Acronym: PENTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB 2013/044/C
Record Dates: First submitted 2013-06-20; First posted 2013-06-27 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol (Active Comparator): Tramadol HCL. Dosage form: Injection Strength: 50mg/ampoule Frequency: 1 time
  Interventions: Drug: Tramadol Injection
- Penthrox (Experimental): Dosage form: Inhalation; Strength: 3ml/bottle; Frequency: Up to 6ml per day. Total weekly dose should not exceed 15ml.
  Interventions: Drug: Penthrox Inhaler

INTERVENTIONS:
Drug: Penthrox Inhaler
  Arms: Penthrox
Drug: Tramadol Injection
  Arms: Tramadol

SUMMARY:
Introduction

Current practice in Singapore Emergency Ambulance Service (EAS) includes the use of analgesia delivered via inhalation Enthanox (Nitrous Oxide). However there are difficulties administering Enthanox on-scene due to the added weight of carrying bulky cylinder tanks. It is common for a delay in administration of analgesia. Inhaled methoxyflurane (Penthrox) is a potential agent for early administration of analgesia by Singapore Civil Defense Force (SCDF) EAS. It is extensively used in the pre-hospital setting in Australia. However data on its use as an analgesic agent in general are limited and there are few published controlled trials of methoxyflurane in an analgesic role. Intramuscular (IM) tramadol is a common medication used in the hospital setting for analgesia. It is well proven, simple to deliver and is not a controlled drug.

Aim

To compare Penthrox and Tramadol in the treatment of acute pain in patients transported by the SCDF EAS.

Methodology

The trial will recruit 400 eligible patients over 1 year (200 Penthrox and 200 tramadol). Patients managed by SCDF EAS for treatment of acute pain and who meet the eligibility criteria will be recruited into the study. Half of SCDF's 30 ambulances (15 ambulances), will be randomly assigned, equipped and trained to carry the new medication (Penthrox). The other half (15 ambulances), will be trained and equipped with tramadol. Allocation will be on a per station level. After 6 months, they will cross over to Penthrox and tramadol respectively.

All paramedics will be trained to use both medications, pain scales and Ramsey scores, and will record patient's pain, sedation scores and patient satisfaction as part of routine clinical practice. All patients will be followed up by a review of their Emergency Department and hospital records for any medication related adverse effects.

Hypothesis

The investigators hypothesize that in patients with acute pain (pain score ≥3), presenting to the ambulance service with musculo-skeletal trauma (limbs or back); pain relief by inhaled methoxyflurane will be equivalent to IM tramadol, as assessed by Visual Analogue Scale (VAS) at 5, 10, 15 and 20 min after start of the study treatments.

DETAILED DESCRIPTION:
Introduction

Current practice in Singapore Emergency Ambulance Service (EAS) includes the use of analgesia delivered via inhalation Enthanox (Nitrous Oxide). However there are difficulties administering Enthanox on-scene due to the added weight of carrying bulky cylinder tanks. It is common for a delay in administration of analgesia. In addition, there are problems with storage, leakage, maintenance and occupational exposure of the EAS crew members. Therefore, there is a need for better standard of care treatment.

Inhaled methoxyflurane (Penthrox) is a potential agent for early administration of analgesia by EAS. It is extensively used in the pre-hospital setting in Australia. However data on its use as an analgesic agent in general are limited and there are few published controlled trials of methoxyflurane in an analgesic role. Intramuscular (IM) tramadol is a common medication used in the hospital setting for analgesia. It is well proven, simple to deliver and is not a controlled drug. We intend to conduct a clinical evaluation trial comparing the use of inhaled Penthrox with IM Tramadol for early pain relief.

Objective & Hypothesis

Primary objectives:

To compare Penthrox (methoxyflurane) and Tramadol in the treatment of acute pain in patients transported by the Singapore Civil Defense Force (SCDF) EAS with respect to:

* Pain Score assessed by Visual Analogue Scale (VAS) at 5,10, 15 and 20 min after start of the study treatment
* Time arrived at scene to delivery of first analgesia
* Time to onset of analgesia (arrive at scene to ≥ 3 point reduction in pain score assessed by VAS)

Secondary Objective:

* To understand patients' perception of pain, satisfaction in pain management, and the use of the analgesic inhaler compared with IM tramadol in the treatment of acute pain.
* To understand staff satisfaction with pain management, and the ease of use of the analgesic inhaler compared with IM tramadol in the treatment of acute pain.
* To assess Ramsay sedation scores at 5, 10, 15 and 20 min after start of the study treatment
* Vital signs (i.e. Respiratory rate, heart rate, blood pressure and GCS)

Methods Study Design

A phased, prospective, non-randomised, before-after evaluation study comparing Penthrox (Methoxyflurane) and Tramadol in patients with acute pain managed by SCDF EAS.

The trial will recruit 400 eligible patients over 1 year (200 Penthrox and 200 tramadol). 200 samples of Penthrox will be provided free of charge by Medical Developments International (MDI), an Australian company, for evaluation during the trial. Patients managed by SCDF EAS for treatment of acute pain and who meet the eligibility criteria will be recruited into the study. Intramuscular tramadol will be purchased by SCDF for this implementation trial.

Half of SCDF's 30 ambulances (15 ambulances), will be randomly assigned, equipped and trained to carry the new medication (Penthrox). The other half (15 ambulances), will be trained and equipped with IM tramadol. Allocation will be on a per station level. After 6 months, the two separate cohort of ambulances will cross over to administer Penthrox and Tramadol and respectively. This is done in order to minimize any potential patient selection bias and ambulance crew operator bias arising in the two 6-monthly time periods.

All paramedics will be trained to use both medications, the pain scales and Ramsey scores, and will record patient's pain, sedation scores patient and staff satisfaction as part of routine clinical practice. In the case when one or both study drugs are used up before the cross-over period, or the patient is ineligible for either drug, SCDF ambulances will still carry Enthanox as a back up analgesia.

SGH will be submitting an ethics application to Centralised Institutional Review Board (CIRB) on behalf of SCDF to recruit all cases presenting to SCDF, irrespective of destination hospital. This is because SCDF does not have its own IRB. All patients will be followed up by a review of their Emergency Department and hospital records for any medication related adverse effects.

Enrollment of Patients Patients will be given the treatment if all eligibility criteria are met and treatment is indicated by protocol. For patients who do not meet inclusion and exclusion criteria for either of the new treatments, Enthanox will still be kept on ambulances during the study period for back up analgesia. No written consent will be sought as this will be part of routine clinical care.

Team members Contribution SCDF staff members will be enrolling eligible participants and administer the study drugs. The SGH study team will provide clinical input into protocols, physician oversight, training for paramedics, data quality control, analysis of data and interpretation of results etc.

Quality Assurance

This study will include the following specific elements for quality assurance:

* Development of standard protocols to perform all data collection and follow-up activities
* Development and adherence to a detailed Standard Operation Procedures (SOP)
* Use of standardized forms and uniform criteria for patient recruitment
* Standardized data processing, editing and generation of edit statements
* Regular communications between the study investigators to resolve questions
* Internal and external monitoring of data collection

Additional steps to ensure data quality include: range checks and verification built into the data entry system and a sequence of logic checking and examination of variables.

Human Subjects Instructions

Risk Reduction

- A formal education and training program will be conducted for all paramedics who will be administering both treatments to patients. This will include didactic and practical training sessions, and competency certification before they will be allow to administer the treatment. Paramedics will also be taught how to monitor patients, watch for adverse effects and how to treat them.

A formal education and training program will be conducted for all investigators who will be conducting surveys to reduce the risks regarding confidentiality. All subjects' identifiers will be removed from the database to protect subjects' confidentiality.

Risk/Benefit

* Comparison of Penthrox and Tramadol will help to advise which drug can be used as a standard drug in the EAS for treatment of acute pain patients. This study has the potential to change practice in Singapore and beyond, and allow patients earlier relief of pain and suffering.

Compensation Plan - No compensation will be provided to the patients or any family members.

Informed Consent Issues

- Apply for waiver of consent for this study. Only collecting patients' pain scale information from SCDF EAS. Therefore, it poses no additional risks to the patients. All patient identifiers will be subsequently removed from the dataset.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pain, with pain score greater than 3, presenting with musculo-skeletal trauma (limbs or back) pain are eligible
* Conscious, haemodynamically stable condition (BP greater than 90/60)
* Age more than 16 years old

Exclusion Criteria:

General

* Females who are nursing or with a positive pregnancy test (pregnant)
* Patients with major head injury or impaired consciousness
* Acute intoxication with drugs or alcohol, or other conditions that might impair ability to score pain
* Chronic pain requiring ongoing use of analgesics
* Abdominal or chest pain (for the purpose of this initial implementation study)

Penthrox only

* Known pre-existing renal or hepatic impairment
* Hypersensitivity to fluorinated anaesthetics or a history of possible adverse reactions in either the patients or relatives (malignant hyperthermia)
* Concomitant use of nephrotoxic medications such as gentamicin or tetracycline

Tramadol only

* Any allergies to tramadol or codeine
* Any history of seizures, epilepsy
* Patients who are taking anti-depressants

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score assessed by Visual Analogue Scale (VAS) | 5, 10, 15 and 20 min

SECONDARY OUTCOMES:
Change in Ramsay sedation Scores | 5, 10, 15 and 20 min

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Civil Defence Force, Singapore, Singapore